CLINICAL TRIAL: NCT02577315
Title: An Open-label, Randomised, Single-dose, Two-way Crossover Study in Healthy Male and Female Subjects to Evaluate the Bioequivalence of Two Fixed Dose Combination Tablets of Empagliflozin 12.5 mg and Metformin 500 mg Compared With the Free Combination of Empagliflozin 25 mg and Metformin 1000 mg Tablets Under Fed Conditions
Brief Title: Demonstrate Bioequivalence of Two 12.5 mg Empagliflozin/500 mg Metformin Fixed Dose Combination Tablets With Free Combination of Empagliflozin 25 mg and Metformin 1000 mg in Healthy Male and Female Volunteers Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1276.27
Record Dates: First submitted 2015-10-08; First posted 2015-10-16 (Estimated); Results first posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin; Metformin

ARMS (2):
- Test - Empagliflozin/Metformin (Experimental): fixed dose combination of 2 tablets of 12.5 mg Empagliflozin and 500 mg Metformin, oral with 200 mL of water uder fed conditions
  Interventions: Drug: Empagliflozin; Drug: Metformin
- Reference - Empagliflozin + Metformin (Experimental): free combination of 1 tablet of 25 mg Empagliflozin and 1 tablet of 1000 mg of Metformin, oral with 200 mL of water under fed conditions
  Interventions: Drug: Empagliflozin; Drug: Metformin

INTERVENTIONS:
Drug: Empagliflozin — Test Therapy - fixed dose combination of 2 tablets of 12.5 mg Empagliflozin and 500 mg Metformin
  Arms: Test - Empagliflozin/Metformin
Drug: Metformin — Test Therapy - fixed dose combination of 2 tablets of 12.5 mg Empagliflozin and 500 mg Metformin
  Arms: Test - Empagliflozin/Metformin
Drug: Empagliflozin — Reference Therapy - free combination of 1 tablets of 25 mg Empagliflozin and 1000 mg Metformin
  Arms: Reference - Empagliflozin + Metformin
Drug: Metformin — Reference Therapy - free combination of 1 tablets of 25 mg Empagliflozin and 1000 mg Metformin
  Arms: Reference - Empagliflozin + Metformin

SUMMARY:
Bioequivalence of two 12.5 mg empagliflozin/500 mg metformin fixed dose combination tablets compared to the free combination of empagliflozin 25 mg and metformin 1000 mg in healthy male and female volunteers under fed conditions

ELIGIBILITY:
Inclusion criteria:

* Healthy male and female subjects aged 18 to 45 years and BMI 18.50 to 24.99 kg/m2 by Quetelet
* Signed informed consent prior to admission to the study
* Subjects must be able to undergo all trial related requests and procedures and follow any trial related restrictions on concomitant medications, diet and life style
* Subjects must be never-smokers or ex-smokers who stopped smoking prior to enrolment (Visit 1)
* Male or female subjects using adequate contraception from at least 30 days before the first study drug administration and until 30 days after trial completion

Exclusion criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and any laboratory value outside the reference range
* Positive results of blood tests for infections (HIV, Syphilis, Hepatitis B or C), urine drug screening test and alcohol breath test
* Any evidence of a concomitant disease judged clinically relevant by the investigator and presence of cardiovascular, respiratory, nervous, endocrine, reproductive, hematopoietic, immune system disorders; gastrointestinal, hepatic, urinary tract, hepatobiliary disorder, mental disturbance
* Surgery of the gastrointestinal tract that could interfere with kinetics of the study drugs (except appendectomy)
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Relevant chronic or aAcute infections/ acute diseases occurred within 4 weeks before inclusion into the study
* History of relevant allergy/hypersensitivity (including allergy to the trial medication or its excipients)
* Regular use of medicinal products less than 2 weeks before investigational drug administration
* Intake of systemic inhibitors or inductors of microsomal hepatic enzymes in less than 30 days before investigational drug administration
* Intake of drugs with a long half-life (¿24 hours) within 30 days or less than 10 half-lives of the respective drug prior to administration of trial medication
* Use of drugs which might reasonably influence the results of the trial based on current knowledge within 14 days prior to drug administration or during the trial
* Participation in another trial with investigational drug administration within 3 months prior to administration of trial medication
* Alcohol intake = 10 units of alcohol per week (1 unit of alcohol equals one 50 ml single measure of distilled alcoholic beverages/spirits (ABV 40%), or 0.5 litre of beer (ABV 5%), or 200 ml glass or red wine (ABV 12%) or history of alcohol abuse, narcomania, or other drug abuse.
* Drug abuse
* Blood donation (more than 100 mL within 30 days prior to administration of trial medication or intended during the trial)
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen as per protocol and per protocol procedures
* Subject is assessed by the investigator as unsuitable for inclusion, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Intake of xanthine-containing drinks or foods and alcohol from 72 h before screening and second treatment period
* Intake of drinks or foods containing grapefruits, Chinese grapefruits, Seville oranges for female subjects:
* Positive pregnancy test, pregnancy or plans to become pregnant within 30 days after study completion
* Breast feeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2015-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1276.27.001 Boehringer Ingelheim Investigational Site, Saint Petersburg, Russia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Actual number of subjects enrolled in fact represents entered / randomized subjects due to the study set up.
Groups:
- Fixed Dose Combination (FDC) / Empagliflozin + Metformin: Participants first received 2 film-coated tablets of 12.5 milligram (mg) Empagliflozin and 500 mg Metformin as a single dose in a fixed dose combination (FDC), then they received free combination of 1 film-coated tablet of 25 mg Empagliflozin and 1 film-coated tablet of 1000 mg Metformin (brand name: Glucophage) as a single dose. The study medication was administered orally in the morning with 200 mL of water after intake of a high-fat, high-caloric meal. Single dose in each treatment period was separated by a washout phase of at least 5 days between drug administrations.
- Empagliflozin + Metformin / Fixed Dose Combination (FDC): Participants first received free combination of 1 film-coated tablet of 25 mg Empagliflozin and 1 film-coated tablet of 1000 mg Metformin (brand name: Glucophage) as a single dose, then they received 2 film-coated tablets of 12.5 milligram (mg) Empagliflozin and 500 mg Metformin as a single dose in a fixed dose combination (FDC). The study medication was administered orally in the morning with 200 mL of water after intake of a high-fat, high-caloric meal. Single dose in each treatment period was separated by a washout phase of at least 5 days between drug administrations.
Period: Treatment Period 1 (4 Days)
Arm/Group | Fixed Dose Combination (FDC) / Empagliflozin + Metformin | Empagliflozin + Metformin / Fixed Dose Combination (FDC)
Started | 12 | 13
Completed | 12 | 12
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout Period (5 Days)
Arm/Group | Fixed Dose Combination (FDC) / Empagliflozin + Metformin | Empagliflozin + Metformin / Fixed Dose Combination (FDC)
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Treatment Period 2 (4 Days)
Arm/Group | Fixed Dose Combination (FDC) / Empagliflozin + Metformin | Empagliflozin + Metformin / Fixed Dose Combination (FDC)
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): all subjects who were randomised to study medication and were documented to have received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fixed Dose Combination (FDC) / Empagliflozin + Metformin | Empagliflozin + Metformin / Fixed Dose Combination (FDC) | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.7 (3.6) | 30.4 (7.8) | 27.6 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13
  Male | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of the Empagliflozin in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of the Empagliflozin in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz). Geometric means (gMeans) represent adjusted gMeans and geometric coefficient of variation (gCV) reflects the intra-individual gCV (%) from the mixed model analysis.
Time Frame: PK plasma samples were taken at: 2 hours (h) before drug administration and 20 minutes, 40 minutes, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 34h, 48h, 72h after drug administration.
Population: Pharmacokinetic analysis set (PKS): all subjects from treated set (TS) who provided at least 1 primary or secondary Pharmacokinetic (PK) endpoint value that was judged as PK evaluable and was not affected by protocol violations relevant to the statistical evaluation. Subject was included, even if he/she contributed only 1 PK value for one period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol (nmol)* hours (h) / Litre (L)
Groups:
- Empagliflozin / Metformin (FDC): Participants received 2 film-coated tablets of 12.5 milligram (mg) Empagliflozin and 500 mg Metformin as a single dose in a fixed dose combination (FDC). The study medication was administered orally in the morning with 200 mL of water after intake of a high-fat, high-caloric meal.
- Empagliflozin + Metformin Free Combination: Participants received free combination of 1 film-coated tablet of 25 mg Empagliflozin and 1 film-coated tablet of 1000 mg Metformin (brand name: Glucophage) as a single dose. The study medication was administered orally in the morning with 200 mL of water after intake of a high-fat, high-caloric meal.
Arm/Group | Empagliflozin / Metformin (FDC) | Empagliflozin + Metformin Free Combination
Number analyzed (Participants) | 24 | 24
nanomol (nmol)* hours (h) / Litre (L) | 6147 (5.4) | 6141 (5.4)
Statistical Analysis 1: Comparison: Empagliflozin / Metformin (FDC) vs Empagliflozin + Metformin Free Combination; Empagliflozin / Metformin (FDC) vs. Empagliflozin + Metformin free combination; Test type: Non-Inferiority or Equivalence — Assessment of bioequivalence was based upon 2-sided 90% confidence intervals (CIs) for the ratio of the geometric means (gMeans) with acceptance range of 80.00 to 125.00%; ANOVA; Analysis of variance (ANOVA) on log scale was used with subjects within sequences as random, whereas sequence, period and treatment as fixed effects; Ratio of geometric means = 100.10, 90% CI 2-sided [97.466 to 102.804] — Relative bioavailability of Empagliflozin was estimated by the ratios of the adjusted geometric means (gMean)

2. Primary Outcome: Area Under the Concentration-time Curve of the Metformin in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of the Metformin in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz). Geometric means (gMeans) represent adjusted gMeans and geometric coefficient of variation (gCV) reflects the intra-individual gCV (%) from the mixed model analysis.
Time Frame: as for outcome 1
Population: Pharmacokinetic analysis set (PKS): all subjects from the TS who provided at least 1 primary or secondary Pharmacokinetic (PK) endpoint value that was judged as PK evaluable and was not affected by protocol violations relevant to the statistical evaluation. Thus, subject was included, even if he/she contributed only 1 PK value for one period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram (ng)*h /millilitre (mL)
Arm/Group | Empagliflozin / Metformin (FDC) | Empagliflozin + Metformin Free Combination
Number analyzed (Participants) | 24 | 24
nanogram (ng)*h /millilitre (mL) | 11912 (13.6) | 12472 (13.6)
Statistical Analysis 1: Comparison: Empagliflozin / Metformin (FDC) vs Empagliflozin + Metformin Free Combination; Empagliflozin / Metformin (FDC) vs. Empagliflozin + Metformin free combination; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 95.51, 90% CI 2-sided [89.29 to 102.16] — Relative bioavailability of Metformin was estimated by the ratios of the adjusted geometric means (gMean)

3. Primary Outcome: Maximum Measured Concentration of the Empagliflozin in Plasma (Cmax)
Description: Maximum measured concentration of the Empagliflozin in plasma (Cmax). Geometric means (gMeans) represent adjusted gMeans and geometric coefficient of variation (gCV) reflects the intra-individual gCV (%) from the mixed model analysis.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Empagliflozin / Metformin (FDC) | Empagliflozin + Metformin Free Combination
Number analyzed (Participants) | 24 | 24
nmol/L | 660 (10.9) | 642 (10.9)
Statistical Analysis 1: Comparison: Empagliflozin / Metformin (FDC) vs Empagliflozin + Metformin Free Combination; Empagliflozin / Metformin (FDC) vs. Empagliflozin + Metformin free combination; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 102.71, 90% CI 2-sided [97.309 to 108.413] — Relative bioavailability of Empagliflozin was estimated by the ratios of the adjusted geometric means (gMean)

4. Primary Outcome: Maximum Measured Concentration of the Metformin in Plasma (Cmax)
Description: Maximum measured concentration of the Metformin in plasma (Cmax). Geometric means (gMeans) represent adjusted gMeans and geometric coefficient of variation (gCV) reflects the intra-individual gCV (%) from the mixed model analysis.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Empagliflozin / Metformin (FDC) | Empagliflozin + Metformin Free Combination
Number analyzed (Participants) | 24 | 24
ng/mL | 1452 (11.3) | 1437 (11.3)
Statistical Analysis 1: Comparison: Empagliflozin / Metformin (FDC) vs Empagliflozin + Metformin Free Combination; Empagliflozin / Metformin (FDC) vs. Empagliflozin + Metformin free combination; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 101.07, 90% CI 2-sided [95.565 to 106.902] — Relative bioavailability of Metformin was estimated by the ratios of the adjusted geometric means (gMean)

5. Secondary Outcome: Area Under the Concentration-time Curve of the Empagliflozin in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC 0-infinity)
Description: Area under the concentration-time curve of the Empagliflozin in plasma over the time interval from 0 extrapolated to infinity (AUC 0-infinity observed). Geometric means (gMeans) represent adjusted gMeans and geometric coefficient of variation (gCV) reflects the intra-individual gCV (%) from the mixed model analysis.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empagliflozin / Metformin (FDC) | Empagliflozin + Metformin Free Combination
Number analyzed (Participants) | 24 | 24
nmol*h/L | 6280 (5.7) | 6261 (5.7)
Statistical Analysis 1: Comparison: Empagliflozin / Metformin (FDC) vs Empagliflozin + Metformin Free Combination; Empagliflozin / Metformin (FDC) vs. Empagliflozin + Metformin free combination; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 100.30, 90% CI 2-sided [97.532 to 103.149] — Relative bioavailability of Empagliflozin was estimated by the ratios of the adjusted geometric means (gMean)

6. Secondary Outcome: Area Under the Concentration-time Curve of the Metformin in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC 0-infinity)
Description: Area under the concentration-time curve of the Metformin in plasma over the time interval from 0 extrapolated to infinity (AUC 0-infinity observed). Geometric means (gMeans) represent adjusted gMeans and geometric coefficient of variation (gCV) reflects the intra-individual gCV (%) from the mixed model analysis.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Empagliflozin / Metformin (FDC) | Empagliflozin + Metformin Free Combination
Number analyzed (Participants) | 24 | 24
ng*h/mL | 12428 (24.8) | 13285 (24.8)
Statistical Analysis 1: Comparison: Empagliflozin / Metformin (FDC) vs Empagliflozin + Metformin Free Combination; Empagliflozin / Metformin (FDC) vs. Empagliflozin + Metformin free combination; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 93.55, 90% CI 2-sided [82.86 to 105.61] — Relative bioavailability of Metformin was estimated by the ratios of the adjusted geometric means (gMean)

ADVERSE EVENTS:
Time Frame: From first drug administration until 14 days after the last drug administration, up to 27 days.
Arm/Group | Empagliflozin / Metformin (FDC) | Empagliflozin + Metformin Free Combination
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 0/24 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.